CLINICAL TRIAL: NCT03864211
Title: Phase I/II Study of Thermal Ablation Followed by Toripalimab in Unresectable Hepatocellular Carcinoma
Brief Title: Thermal Ablation Followed by Immunotherapy for HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RI11330
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; Immunotherapy; Thermal ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Transurethral Resection of Prostate; toripalimab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toripalimab monotherapy (Active Comparator): Toripalimab is administrated intravenously (240mg, Q3W) continuously until documented disease progression, discontinuation due to toxicity withdrawal of consent or the study ends.
  Interventions: Drug: Toripalimab
- Thermal ablation plus toripalimab (Experimental): One to five target lesions will be ablated completely. Toripalimab therapy will be initiated on day 3 or day 14 after ablation ((240mg, Q3W) ). Toripalimab is administrated continuously until documented disease progression, discontinuation due to toxicity withdrawal of consent or the study ends.
  Interventions: Procedure: Thermal ablation; Drug: Toripalimab

INTERVENTIONS:
Procedure: Thermal ablation — Radiofrequency ablation or microwave ablation is performed under CT or ultrasound guidance for one to five target lesions.
  Arms: Thermal ablation plus toripalimab
Drug: Toripalimab — Protocol 1. Patients received toripalimab (240mg, Q3W) as monotherapy.
  Protocol 2. Patients received toripalimab (240mg, Q3W) on day 3 after ablation.
  Protocol 3. Patients received toripalimab (240mg, Q3W) on day 14 after ablation.
  Other Names: Immunotherapy

SUMMARY:
The purpose of this study is to determine the safety and efficacy of immunotherapy toripalimab (anti-PD-1 mAb) combined with thermal ablation in patients with Hepatocellular Carcinoma (HCC).

DETAILED DESCRIPTION:
1.1 Primary Objective & Hypothesis Determine the safety and efficacy of radiofrequency ablation (RFA)/microwave ablation (MWA) followed by toripalimab for advanced HCC by establishing the rates of toxicity that occur within 6 months after ablation. Hypothesis: Thermal ablation followed by toripalimab will have similar toxicity to toripalimab monotherapy. Thermal ablation enhances antitumor immune response and improves the best overall response rate compared to historical controls with toripalimab alone.

1.2 Secondary Objectives and Hypotheses Estimate the progression-free survival, and overall survival. Hypothesis: Disease control and survival will be better than that observed with toripalimab monotherapy.

1.3 Exploratory Objectives Explore changes in inflammatory biomarkers (including, but not limited to CD8+/Treg ratio, total CD4+ counts, total lymphocyte count) in pretreatment and on-treatment serially collected peripheral blood samples. Hypothesis: Changes in inflammatory biomarkers after thermal ablation may correlate with a more favorable response to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* With hepatocellular carcinoma, who meet the clinical diagnostic criteria of Primary HCC confirmed by histopathology, cannot undergo radical resection or radical ablation, and fail or intolerable to first-line systemic therapy
* Be willing and able to provide written informed consent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have ECOG performance status 0-1.
* Pretreatment CT chest /abdomen /pelvis within 14 days of protocol enrollment.
* Pathologic diagnosis of hepatocellular carcinoma (including fibrolamellar variants and biphenotypic tumors with a HCC component).
* Child Pugh Class A or B (score =7)
* Deemed ineligible for curative intent therapy with surgical resection or locoregional treatment or that had progression with at least 3 lesions thereafter.
* At least one lesion can be completely ablated by radiofrequency/microwave ablation.
* The the maximum diameter of a single lesion is less than 10 cm. Tumors account for less than 50% of the liver volume.
* Patients with extrahepatic disease are eligible.
* Progress or intolerance following at least one systemic treatment regimen.
* Have measurable disease based on RECIST 1.1.
* Demonstrate adequate organ function. Adequate Organ Function Laboratory Values System Laboratory Value Hematological Platelets ≥ 50,000 /mL Hepatic Serum total bilirubin ≤ 3 mg/dL AST (SGOT) and ALT (SGPT) ≤ 5 X ULN.
* Subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 150 days after the last dose of study therapy (for women of child-bearing potential) or 210 days after the last dose of study therapy (for men who have partners of child-bearing potential).
* Have a life expectancy of greater than 3 months (in the opinion of the treating physician).

Exclusion Criteria:

* Received local ablation or external beam radiation within 3 months .
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose of >10 mg prednisone daily or equivalent at time of first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a known additional malignancy that is progressing or requires active treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with allografts (including liver transplants) are not eligible for this protocol.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has received a live vaccine within 30 days of planned start of study therapy.
* Prior anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA4 immunotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Up to approximately 3 years
  From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall response rate | Up to approximately 2 years
  Treatment evaluation will be done using mRECIST
Overall survival | Up to approximately 3 years
  From random date to death for any reason.
Disease Control Rate | Up to approximately 3 years
  Defined as the percentage of patients who have achieved complete response, partial response and stable disease
Number of participants with adverse events | Up to approximately 3 years
  Evaluation will be done using NCI-CTCAE (version 4.03).
Tumour marker response | Up to approximately 3 years
  Percentage of AFP variation
The time to deterioration of quality of life | Up to approximately 3 years
  Repetitive decreases of 10 points or more from the baseline of the EORTC QLQ-C30 for two consecutive assessments or a decrease of 10 points or more in a single assessment followed by death from any cause within three weeks.
Duration of response | Up to approximately 2 years
  the time from first documented complete or partial response to disease progression or death) according to investigator-assessed and independently-assessed mRECIST criteria
The general health status | Up to approximately3 years
  The Eastern Cooperative Oncology Group (ECOG) was applied to assess the general health status of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Liangrong Shi, M.D., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Shi L, Chen L, Wu C, Zhu Y, Xu B, Zheng X, Sun M, Wen W, Dai X, Yang M, Lv Q, Lu B, Jiang J. PD-1 Blockade Boosts Radiofrequency Ablation-Elicited Adaptive Immune Responses against Tumor. Clin Cancer Res. 2016 Mar 1;22(5):1173-1184. doi: 10.1158/1078-0432.CCR-15-1352. PMID 26933175
- [Background] Chu KF, Dupuy DE. Thermal ablation of tumours: biological mechanisms and advances in therapy. Nat Rev Cancer. 2014 Mar;14(3):199-208. doi: 10.1038/nrc3672. PMID 24561446
- [Background] Ulahannan SV, Duffy AG. Hepatocellular carcinoma and immune therapy, from a clinical perspective; where are we? Hepat Oncol. 2016 Aug;3(3):183-185. doi: 10.2217/hep-2016-0008. Epub 2016 Aug 19. No abstract available. PMID 30191038
- [Background] Keam SJ. Toripalimab: First Global Approval. Drugs. 2019 Apr;79(5):573-578. doi: 10.1007/s40265-019-01076-2. PMID 30805896
- [Background] Hwang WL, Pike LRG, Royce TJ, Mahal BA, Loeffler JS. Safety of combining radiotherapy with immune-checkpoint inhibition. Nat Rev Clin Oncol. 2018 Aug;15(8):477-494. doi: 10.1038/s41571-018-0046-7. PMID 29872177
- [Background] Taube JM, Klein A, Brahmer JR, Xu H, Pan X, Kim JH, Chen L, Pardoll DM, Topalian SL, Anders RA. Association of PD-1, PD-1 ligands, and other features of the tumor immune microenvironment with response to anti-PD-1 therapy. Clin Cancer Res. 2014 Oct 1;20(19):5064-74. doi: 10.1158/1078-0432.CCR-13-3271. Epub 2014 Apr 8. PMID 24714771